CLINICAL TRIAL: NCT07218133
Title: Trans-Auricular Stimulation for Postoperative Inflammation in Spine Surgery
Brief Title: Auricular Vagal Nerve Stimulation for Spinal Fusion Surgery
Acronym: TAPIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander T. Yahanda (Other)
Responsible Party: Sponsor-Investigator, Alexander T. Yahanda, Neurosurgery Resident, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202407057SpineVNS
Record Dates: First submitted 2025-10-08; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Spinal Fusion; Hyperglycemia; Postoperative Pain Management; Postoperative Care; Spine Disease; Neurologic Deficits; Neurological Disorder; Inflammation; Spine Condition; Spinal (Fusion) Surgery; Cytokine Levels; Spine Fusion
Keywords: spinal fusion; postoperative pain; glycemic control; inflammation; vagal nerve stimulation; postoperative complications; cytokine; spine surgery
MeSH Terms: conditions — Hyperglycemia; Spinal Diseases; Neurologic Manifestations; Nervous System Diseases; Inflammation; Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the vagal nerve stimulation arm or the sham stimulation arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be fitted with an auricular stimulator, but blinded to whether they are receiving stimulation or not. Outcome scores will be assessed and recorded by clinicians blinded to treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Auricular vagal nerve stimulation (Experimental): Participants will receive vagal nerve stimulation twice on the day of surgery (once preoperatively) and twice daily postoperatively for duration of hospitalization.
  All patients will be fitted with the device via adhesive contacts to the left ear. Stimulation will occur for 20 minutes per session. The intervention will provide stimulation according to the following parameters: frequency 20 Hz, pulse width 250 µm, and fixed intensity of 0.5 milliampere. The amplitude of stimulation may be reduced if a patient complains of discomfort at the site of stimulation
  Interventions: Device: Auricular vagus nerve stimulation
- Sham vagal nerve stimulation (Sham Comparator): Participants will have an auricular vagal nerve stimulator device applied in the same manner as the experimental arm, but they will not receive the actual stimulation.
  Interventions: Device: Sham Auricular Vagus nerve Stimulation

INTERVENTIONS:
Device: Auricular vagus nerve stimulation — Transcutaneous auricular vagal nerve stimulation
  Arms: Auricular vagal nerve stimulation
Device: Sham Auricular Vagus nerve Stimulation — Transcutaneous auricular vagal nerve stimulator applied without utilizing stimulating current.
  Arms: Sham vagal nerve stimulation

SUMMARY:
This study is a randomized controlled trial that will evaluate the effect of non-invasive auricular vagal nerve stimulation on inflammatory markers, glycemic control, postoperative pain, and inflammation-related clinical outcomes after long-segment spinal fusion surgeries when compared to current accepted management.

DETAILED DESCRIPTION:
Long-segment spinal fusions are effective interventions to relieve pain, neurological compromise, or disability related to a variety of causes of advanced spinal degeneration or spinal deformity. Despite advancements in minimally invasive spine surgery, revision of prior instrumentation, correction of coronal or sagittal imbalance, bony decompression, and multilevel arthrodesis often must be performed via open surgery. While these procedures can produce excellent results with regards to postoperative alignment, neural decompression, and functional improvement, they are long and invasive cases requiring large incisions and extensive soft tissue dissection and osseous manipulation. As such, postoperative adverse events or complications are common (e.g., DVT/PE, wound healing problems, infection, nerve stretch injury, etc.). These patients almost universally experience significant postoperative pain, require postoperative rehabilitation, and are at high-risk for hospital readmissions. Moreover, the sterile trauma from long-segment spinal surgeries is a tremendous systemic inflammatory stimulus that yields downstream sequelae such as hyperglycemia, elevated inflammatory markers (e.g. cytokines), signs of microvascular ischemia, and other stress-related outcomes. Attempts to control this inflammation and reduce the adverse effects of these surgeries are lacking, particularly with respect to non-pharmacologic options.

Vagal nerve stimulation (VNS) is a promising emerging modality by which the body's systemic inflammatory response may be attenuated. Importantly, VNS may be successfully applied via noninvasive auricular stimulation. This technique has been trialed as non-pharmacologic pain control adjunct after multiple types of surgeries or painful medical events, but none as traumatic as long-segment spinal fusion. It also has been shown to yield substantial anti-inflammatory effects in numerous animal models. Furthermore, auricular VNS has been extensively studied at Washington University School of Medicine in multiple neurological conditions, including aneurysmal subarachnoid hemorrhage, acute ischemic stroke, and intraparenchymal hemorrhage. The use of noninvasive VNS devices has been shown to be an intervention that is safely administered and does not cause undue distress to patients. Given these promising aspects of VNS, Washington University's particular interest in this treatment modality, and the unmet postoperative care needs for long-segment spinal fusion patients, the investigators propose prospectively studying the effects of auricular VNS in a population of patients at Barnes-Jewish Hospital who have undergone long-segment fusion surgeries. The investigators hypothesize that perioperative VNS will mitigate the systemic inflammatory reaction in these patients as demonstrated by reduced inflammatory markers (both direct and indirect) and improved inflammatory-mediated clinical outcomes.

This study will be a randomized controlled trial assessing differences between accepted perioperative care plus auricular VNS (the intervention) as compared to accepted perioperative care plus a sham stimulus. The VNS device will be a noninvasive stimulator applied to the left ear to stimulate the auricular branch of the vagus nerve. All patients will be fitted with the device, and the sham stimulus will not receive the required therapeutic stimulation through the device. Patients will receive stimulation twice on the day of surgery followed by twice daily during the duration of their postoperative hospital admission. Relevant inflammatory cytokines, laboratory tests, pain scores, clinical outcomes, and imaging studies will be obtained for each patient. Post-hospital disposition, delayed adverse outcomes, and hospital readmissions will also be tracked after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Long-segment spinal fusions (defined as constructs spanning at least L2-pelvis for thoracolumbar fusions or C2-T2 for cervical fusions)
* Ability to undergo a reliable neurologic examination and pain assessments

Exclusion Criteria:

* Patients <18 years of age
* Shorter-segment spinal fusions than those described above
* Undergoing current active cancer therapy
* Undergoing treatment with immunosuppressive drugs
* Additional spinal surgery within past 6 months
* Sustained bradycardia or presence of pacemaker
* History of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokine levels | 5-10 days (depending on hospital admission length)
  The levels of 4 different inflammatory cytokines will be measured: interleukin-6 (IL-6), IL-1, IL-10, and tumor necrosis factor alpha (TNF-a) (all measured in pg/ml). Blood for these tests will be drawn preoperatively, postoperatively, on postop day 3, and postop day 6 (or time of discharge).

SECONDARY OUTCOMES:
Pain scores | 5-10 days (depending on hospital admission length)
  Patient pain levels will be assessed twice daily using the visual analogue scale (VAS), a validated pain reporting scale that uses a 100-millimeter horizontal line with anchors at "no pain" (0) and "worst possible pain" (100). Patients draw a line along this spectrum to signify their pain level. Higher distance along the spectrum in a left-to-right direction indicates higher pain.
blood glucose levels | 5-10 days (depending on hospital admission length)
  Glucose measurements will be obtained multiple times daily via bedside point-of-care testing as well as through daily CMP labs (in mg/dL).
Postoperative adverse events/complications | 5-10 days (depending on hospital admission length)
  Investigators will track the incidence of postoperative adverse events or complications, including temporary radiculopathy or nerve stretch injury, deep vein thrombosis (DVT), pulmonary embolism (PE), acute kidney injury (AKI), ileus, wound healing problems, hospital delirium, transfusion reactions, and infections. All patients will receive screening lower extremity doppler (LED) studies before surgery and at time of hospital discharge.
Secondary markers of inflammation | 5-10 days (depending on hospital admission length)
  Daily laboratory studies that serve as surrogate markers for the body's degree of systemic inflammation will be obtained. This includes labs such as CRP, cortisol, creatinine, and troponin (all in mg/dL)
Post-hospitalization disposition | 5-10 days (depending on hospital admission length)
  Investigators will track patients' post-hospitalization disposition (e.g. home versus inpatient rehabilitation).
Heart rate | Time Frame: 5-10 days (depending on hospital admission length)
  Investigators will continuously monitor patients' heart rates to capture incidences of bradycardia that may be associated with the VNS intervention.
Opioid usage | 5-10 days (depending on hospital admission length)
  Patients' daily opioid usage will be recorded while hospitalized. Usage will be converted to morphine milligram equivalents (MME).
Insulin requirements | 5-10 days (depending on hospital admission length)
  Insulin requirements (units insulin) for patients during their hospital stay will be recorded.
Erythrocyte sedimentation rate (ESR) | 5-10 days (depending on hospital admission length)
  Postoperative ESR will be measured daily (in mm/hr) to assess systemic inflammation.
D-dimer levels | 5-10 days (depending on hospital admission length)]
  D-dimer levels will be obtained postoperatively every other day (in microgram/mL)
Hospital admission length | 5-10 days (depending on hospital admission length)
  Length of patient hospital stay after surgery will be recorded.
Blood pressure | 5-10 days (depending on hospital admission length)]
  Tracking of blood pressure and temperature will allow investigators to evaluate the potential influence of VNS on blood pressure control for hypertensive patients and to determine if any hypotensive events are associated with the intervention.
Readmission rates | 60 days postoperatively
  The incidence of hospital readmission within 30 days and 60 days will be recorded (yes versus no readmissions).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No